CLINICAL TRIAL: NCT00898235
Title: Data, Tissue, Blood, and Urine Repository for Amyloid Diseases
Brief Title: Collection of Samples and Clinical Data From Patients With Amyloid Diseases
Status: Recruiting | Type: Observational
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: H-22838; CDR0000632869 (Other Grant/Funding Number: Amyloid Resarch Fund at BUSM)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis | interventions — Polymerase Chain Reaction; Spectrometry, Fluorescence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, and tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: clonality analysis — analyze clonality
Genetic: polymerase chain reaction — analyze polymerase chain reaction
Genetic: protein analysis — analyze protein
Other: biologic sample preservation procedure — preserve biologic samples
Other: laboratory biomarker analysis — analyze laboratory biomarkers
Procedure: fluorescence spectroscopy — perform fluorescence spectroscopy on specimens
Procedure: quality-of-life assessment — assess quality of life at each follow-up for life

SUMMARY:
RATIONALE: Collecting and storing samples of blood, urine, tissue and data from patients with amyloid diseases to test in the laboratory may help the study of this disease in the future.

PURPOSE: This research study is collecting samples from patients with amyloid diseases

DETAILED DESCRIPTION:
OBJECTIVES:

* To establish and maintain a database of clinical material (i.e., blood, urine, and tissue) and information on patients with amyloid diseases.

OUTLINE: Blood, urine, tissue, and bone marrow samples are collected during standard laboratory evaluations to maintain a repository of biospecimens in the Gerry Amyloid Research Laboratory, to permit the correlation of clinical results with measured biological events, and for future research studies. Bone marrow RNA samples are examined for immunoglobulin light-chain gene sequences and amino acids by polymerase chain reaction and positional cloning. Blood serum and urine samples are evaluated for amyloid protein stability by high-resolution calorimetry, isothermal-titration calorimetry, and far- and near-UV circular dichroism and fluorescence spectroscopy. Urine samples are also examined for post-translational modifications (e.g., glycosylation, sulfation, and cross-linking) to identify common features unique to amyloid proteins. Tissue samples are analyzed for biochemical and biophysical properties and for post-translational modifications in light chains.

Quality of life is assessed by the 36-Item Short Form Survey (SF-36).

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Diagnosis or suspicion of amyloidosis

PATIENT CHARACTERISTICS:

* Referred to the Amyloid Treatment and Research Center at Boston University Medical Center

PRIOR CONCURRENT THERAPY:

* Not specified

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed, or with suspicion of having, amyloidosis
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2000-01 (Actual); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Establish a repository to promote biochemical research | life of study

SECONDARY OUTCOMES:
Collection of clinical material and information | life of study

CONTACTS AND LOCATIONS:
Overall Officials: Vaishali Sanchorawala, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston University Cancer Research Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ramireddy S, Prokaeva T, Chen H, Spencer B, Wong S, Dasari S, Dao L, McPhail ED, Sanchorawala V, Mendelson L. The Amyloidosis Intersection: Dual Amyloid Types in a Single Host. Eur J Haematol. 2025 Sep;115(3):287-298. doi: 10.1111/ejh.14429. Epub 2025 Jun 17. PMID 40526008
- [Derived] Staron A, Burks EJ, Lee JC, Sarosiek S, Sloan JM, Sanchorawala V. Assessment of minimal residual disease using multiparametric flow cytometry in patients with AL amyloidosis. Blood Adv. 2020 Mar 10;4(5):880-884. doi: 10.1182/bloodadvances.2019001331. PMID 32130406
- [Derived] Staron A, Connors LH, Ruberg FL, Mendelson LM, Sanchorawala V. A new era of amyloidosis: the trends at a major US referral centre. Amyloid. 2019 Dec;26(4):192-196. doi: 10.1080/13506129.2019.1640672. Epub 2019 Jul 15. PMID 31306033
- [Derived] Lilleness B, Ruberg FL, Mussinelli R, Doros G, Sanchorawala V. Development and validation of a survival staging system incorporating BNP in patients with light chain amyloidosis. Blood. 2019 Jan 17;133(3):215-223. doi: 10.1182/blood-2018-06-858951. Epub 2018 Oct 17. PMID 30333122
- [Derived] Shu J, Lo S, Phillips M, Sun F, Seldin DC, Berenbaum I, Berk JL, Sanchorawala V. Depression and anxiety in patients with AL amyloidosis as assessed by the SF-36 questionnaire: experience in 1226 patients. Amyloid. 2016 Sep;23(3):188-193. doi: 10.1080/13506129.2016.1208081. Epub 2016 Jul 27. PMID 27460276
- [Derived] Cowan AJ, Skinner M, Seldin DC, Berk JL, Lichtenstein DR, O'Hara CJ, Doros G, Sanchorawala V. Amyloidosis of the gastrointestinal tract: a 13-year, single-center, referral experience. Haematologica. 2013 Jan;98(1):141-6. doi: 10.3324/haematol.2012.068155. Epub 2012 Jun 24. PMID 22733017